CLINICAL TRIAL: NCT04954677
Title: A Prospective Randomized Controlled Trial of AI-box , a Real-time Quality Control System of Magnetic-controlled Capsule Gastroscopy.
Brief Title: A Real-time Quality Control System of Magnetic-controlled Capsule Gastroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Ancon Technologies Ltd (Industry); Shandong Provincial Hospital (Other Government); Binzhou Medical University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice President of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2021-SDU-QILU-087
Record Dates: First submitted 2021-06-18; First posted 2021-07-08 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Magnet Controlled Capsule Endoscopy
Keywords: Artificial intelligence; Deep learning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participates and outcomes Assesors will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participates being subjected to capsule endoscopy (AI-box assistant) (Experimental): In this group ,Participates will be subjected to magnetically controlled capsule gastroscopy with AI-box assistant.
  Interventions: Other: AI-box
- Participates being subjected to capsule endoscopy (No Intervention): In this group ,Participates will be subjected to magnetically controlled capsule gastroscopy without AI-box assistant.

INTERVENTIONS:
Other: AI-box — Automatic quality-control system（AI-box）could real-time measure endoscopic inspection completeness, evaluate gastric cleanliness.
  Arms: Participates being subjected to capsule endoscopy (AI-box assistant)

SUMMARY:
With the rapid development of artificial intelligence technology, more and more deep learning technology has been applied to medicine. Our research is to develop a set of quality control system for magnetic capsule gastroscope using deep learning technology, and conduct a randomized controlled trial to verify its practical efficiency.

DETAILED DESCRIPTION:
The accuracy of magnetic controlled capsule endoscopy(MCCE) in the diagnosis of stomach lesions is highly consistent with the traditional electronic gastroscopy. It has become a new comfortable and safe form for screening and It is also the beneficial complementarity of the traditional electronic gastroscope. To ensure the medical quality of magnetic controlled capsule endoscopy system, Based on Artificial Intelligence Deep Learning Technology ,investigators developed the Magnetic-controlled Capsule Endoscopic Assisted Quality Control System(AI-box).Randomized controlled trials will be conducted on prospective subjects to verify the quality control efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged 18-75 years old who underwent MCCG examination in Qilu Hospital of Shandong University, Shandong Provincial Hospital affilated to Shandong First Medican University, and the Binzhou Medical University Hospital.

Exclusion Criteria:

* People who are allergic to the ingredients prepared in the stomach before examination;
* Patients with astrointestinal bleeding or ulcers, or prior gastrointestinal bleeding or ulcers within the last 24 months;
* Patients with esophageal and gastric tumor diseases that are undergoing active surgical treatment;
* Contraindications to the MCE test, including suspected or known gastrointestinal obstruction, stenosis, fistula, diverticula, etc; presence of gastrointestinal obstruction symptoms such as pain or dysphagia;
* Prior gastrointestinal tract or abdominal surgery other than simple procedures which would not change the gastrointestinal tract anatomy, such as polyp removal, cholecystectomy or appendectomy;
* Inoperative conditions or refusal to undergo abdominal surgery if required (ie, if the capsule will not pass and cannot be removed by endoscopy);
* A cardiac pacemaker is installed in the body, except when the pacemaker is a new MRE-compatible product;
* Electronic devices such as cochlear implant, magnetic metal drug infusion pump, nerve stimulator and magnetic metal foreign body are implanted in vivo;
* Planned MRI examination before capsule endoscopy discharge;
* Pregnant women;
* Patients with deglutition disorders or gastric emptizing disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Mean inspection completeness | 4 months
  After the inspection，investigators will review the whole process of inspection and record the sites observed as well as unobserved sites，then calculate the inspection completeness（number of observed sites in each patient/10）besides the the blind spot rate(number of unobserved sites in each patient/10 ) per procedure in control group and AI-assisted group.

SECONDARY OUTCOMES:
Cleanliness judgement consistency between expert and AI-box | 4 months
  After the inspection，investigators will review the whole process of inspection and make a judgement of cleanliness of different sites of gastric then compared with the cleanliness judgement of AI-box. So at last investigators will calculate the accuracy of the AI result.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China